CLINICAL TRIAL: NCT05869760
Title: Observational Validation of Skin Carotenoid Biomarker of Infant and Toddler Carotenoid Intake
Brief Title: Baylor Infant and Toddler Biomarker of Nutrition Study
Acronym: BITBONS
Status: Recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Houston (Other); East Carolina University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Nancy Engelmann Moran, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-52929; 1R01HD111555 (NIH)
Record Dates: First submitted 2023-05-12; First posted 2023-05-22 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Healthy Nutrition; Healthy Diet
Keywords: infant; toddler; carotenoids; biomarkers; food intake; visual development; contrast sensitivity; skin carotenoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, human milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational Group: Children will be followed from 4-24 months of age.
  Interventions: Other: Carotenoid Intake; Other: Serum carotenoid concentrations

INTERVENTIONS:
Other: Carotenoid Intake — Carotenoid intake calculated from food diary records reported by guardians.
Other: Serum carotenoid concentrations — Serum carotenoid concentrations measured by HPLC.

SUMMARY:
Young children rely on their foods and drinks for the nutrients they need to grow, like energy, protein, vitamins, and minerals. In addition to nutrients, there are substances in fruits, vegetables, milk and formula, called phytochemicals, that can support health. While researchers know more about the role of phytochemicals in adult health, researchers know surprisingly little about how phytochemicals can support health in young children. One group of phytochemicals are called the carotenoids. Carotenoids are responsible for the red, orange, and yellow colors in some fruits and vegetables. In adults, carotenoids can support visual function. Researchers also know that measuring levels of carotenoids in the blood or optically in the skin, can serve as an indirect measurement of what child and adults eat.

The purpose of this study is to determine how a child's usual intake of carotenoids is related to their visual development and their blood and skin levels of carotenoids. The study involves 6 visits. For each visit, we will ask about the child's recent diet, will measure their body size, collect a blood sample, collect optical measurements of their skin, and will test how sharp their vision is.

DETAILED DESCRIPTION:
Early life nutrition is recognized as key determinant of short- and long-term health. However, a lack of objective, reliable, and valid methods to determine what exactly children makes it difficult to carefully study nutrition in infants and toddlers.

Carotenoids are fat-soluble pigments found primarily in fruits and vegetables (F&Vs) that support healthy functioning. Carotenoids support vitamin A requirements, reduce inflammation and cancer risk, and support cognitive, visual, and cardiovascular health. Since carotenoids are colorful, researchers can easily measure them in blood and tissues using color-measuring devices. Blood carotenoid concentrations are used as biomarkers of adult F&V intake. Advances in carotenoid measurement technologies may make carotenoid biomarker measures in children more feasible. However, the precision and accuracy of these biomarkers in children is not as well understood.

With better measures of carotenoid intake comes the opportunity to understand how carotenoid intake relates to children's health. A high priority area to investigate in this young children is whether dietary carotenoids are associated with visual function. Lutein and zeaxanthin, carotenoids that accumulate in the back of the eye (macula), are associated with visual contrast sensitivity in children and adults, a visual function which may support children's interactions with their environments, but this association has not been sufficiently studied in healthy infants and toddlers. In this study, the investigators will define in infants and toddlers 1) the rigorous validation of a skin carotenoid biomarker of dietary intake and 2) the associations between carotenoid intake and visual function.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* born at term (more than or equal to 37 weeks gestation)
* between the 1st to 99th weight for age percentile at 3 months of age
* participating guardian speaks, reads, and understands English
* guardian categorizes child as non-Hispanic white, Hispanic white, Asian, or non-Hispanic Black

Exclusion Criteria:

* physician-diagnosed metabolic, absorptive, or endocrine condition
* diagnosed food intolerance or allergy
* has a sibling enrolled in the study

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy infants and toddlers, born at term, and who are between the 1st and 99th percentile will be enrolled at 3 months of age. Children are categorized by their adult guardian as non-Hispanic white, Hispanic white, Asian, or non-Hispanic Black. Child participants are free of physician diagnosed metabolic, absorptive, or endocrine conditions, do not have diagnosed food intolerances or allergies, and do not have a sibling enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Skin Carotenoid Score-4 months | 4 months of age
  Finger skin carotenoid score measured by pressure-mediated reflection spectroscopy
Skin Carotenoid Score-6 months | 6 months of age
  Finger skin carotenoid score measured by pressure-mediated reflection spectroscopy
Skin Carotenoid Score-8 months | 8 months of age
  Finger skin carotenoid score measured by pressure-mediated reflection spectroscopy
Skin Carotenoid Score-12 months | 12 months of age
  Finger skin carotenoid score measured by pressure-mediated reflection spectroscopy
Skin Carotenoid Score-18 months | 18 months of age
  Finger skin carotenoid score measured by pressure-mediated reflection spectroscopy
Skin Carotenoid Score-24 months | 24 months of age
  Finger skin carotenoid score measured by pressure-mediated reflection spectroscopy

SECONDARY OUTCOMES:
Contrast Sensitivity - 4 months | 4 months of age
  Contrast sensitivity measured by Mayer-Kran Double Happy Test
Contrast Sensitivity - 6 months | 6 months of age
  Contrast sensitivity measured by Mayer-Kran Double Happy Test
Contrast Sensitivity - 8 months | 8 months of age
  Contrast sensitivity measured by Mayer-Kran Double Happy Test
Contrast Sensitivity - 12 months | 12 months of age
  Contrast sensitivity measured by Mayer-Kran Double Happy Test
Contrast Sensitivity - 18 months | 18 months of age
  Contrast sensitivity measured by Mayer-Kran Double Happy Test
Contrast Sensitivity - 24 months | 24 months of age
  Contrast sensitivity measured by Mayer-Kran Double Happy Test

CONTACTS AND LOCATIONS:
Locations (1):
- USDA/ARS Children's Nutrition Research Center, Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided